CLINICAL TRIAL: NCT03994718
Title: Creative Arts Interventions for Improved Epilepsy Patient Quality of Life
Brief Title: Creative Arts II Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Endowment for the Arts, United States (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D19124
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Epilepsy
Keywords: art; music; visual art; writing; epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music (Experimental): The musician will either offer music that can either be played for the participant or an instrument so they can experience playing themselves. The duration of the intervention will be determined by participant interest and tolerance, but not to exceed 60 minutes. The outpatient music intervention will consist of providing a recording of similar music for the participant to listen to for at least 30 minutes per week, along a with telephone call session with the music therapist.
  Interventions: Other: Music intervention
- Visual art (Experimental): The creative visual artist will assess interest in spending time using the materials provided. Participants will be offered watercolor painting, drawing, or adult coloring. There will be a guided activity based on their art making preference. A standardized prompt will be utilized for both writing and visual art sessions. The duration of the intervention will be determined by participant interest and tolerance, but not to exceed 60 minutes. For remote follow-up sessions, participants will be supplied with a small art kit to use at home.
  Interventions: Other: Visual arts intervention
- Creative writing (Experimental): The writer will ask the participant about their interests and experiences in writing or storytelling. The following options are offered; introduction to journaling, storytelling or writing exercises with prompts to get started, interactive writing or storytelling activities. For participants who are unable to write or prefer not to, the writer can scribe their words on a laptop and print them out. The duration of the intervention will be determined by participant interest and tolerance, but not to exceed 60 minutes. For follow-up sessions, participants will be supplied with a journal.
  Interventions: Other: Creative writing intervention

INTERVENTIONS:
Other: Music intervention — The music therapist will work with subjects for up to 60 minutes each session.
  Arms: Music
Other: Visual arts intervention — The visual artist will work with subjects for up to 60 minutes each session.
  Arms: Visual art
Other: Creative writing intervention — The creative writer will work with subjects for up to 60 minutes each session.
  Arms: Creative writing

SUMMARY:
The purpose of this study is to determine the impact of music, visual art, or creative writing on quality of life measures for epilepsy patients.

DETAILED DESCRIPTION:
Qualifying patients admitted to Epilepsy Monitoring Unit will be approached for participation in the study. Patients who consent will be randomly assigned to work with one of three creative artists (visual artist, creative writer, or therapeutic musician. The assigned artist will provide 1 intervention while the patient is admitted and 4 follow-up interventions after discharge from the hospital. Follow-up sessions will be conducted remotely, either by phone or over the internet.

Subjects will be asked to complete study questionnaires before and after the first art intervention, and again after the last follow-up session. The study seeks to measure the impact of arts interventions on quality of life. Secondary objectives include the effects of the interventions on seizure frequency and EEG spike generation, as well as the impact of creative arts interventions on patients diagnosed with non-epileptic events during hospitalization.*

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Scheduled for admission to the Dartmouth-Hitchcock Medical Center Epilepsy Monitoring Unit for diagnostic Video/EEG monitoring
3. Capable of giving informed consent.
4. Able to follow instructions

Exclusion Criteria:

1. Active psychiatric illness that would interfere with participation with the artist.
2. Active general medical condition that would impair the participant's consciousness or ability to participate.
3. Any other reason that, in the opinion of the investigator, would exclude the participant from successful participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in participant Quality of Life (QOLIE-10) scores before and after the interventions. | Each participant will be assessed at baseline (Day 1) and after the inpatient intervention (approximately Day 3 - 21) and at baseline (Day 1) and after the follow-up remote interventions (approximately 8 weeks after discharge).
  Change in quality of life will be calculated using the QOLIE-10 questionnaire responses.The QOLIE-10 includes 10 questions with a total score range of 10 - 51. The score will be calculated by the sum of scores for all questions divided by the number of items answered. Thus, if a patient skipped an item, it is not reflected in the total score. A lower score indicates a higher quality of life, and a higher score indicates a lower quality of life.
Change in participant Distress scores before and after the interventions. | Each participant will be assessed at baseline (Day 1) and after the inpatient intervention (approximately Day 3 - 21) and at baseline (Day 1) and after the follow-up remote interventions (approximately 8 weeks after discharge).
  Change in distress will be calculated using the Distress scale. The Distress scale asks patients to rate their distress on a scale from 0 - 10, with 0 meaning "no distress" and 10 meaning "extreme distress." Lower scores indicate less distress.

SECONDARY OUTCOMES:
Change in participant Patient Health Questionnaire (PHQ-9) scores before and after interventions. | Each participant will be assessed at baseline (Day 1) and after the inpatient intervention (approximately Day 3 - 21) and at baseline (Day 1) and after the follow-up remote interventions (approximately 8 weeks after discharge).
  Change in health status will be calculated using the PHQ-9 questionnaire. The PHQ-9 is a 9-item questionnaire with scores ranging from 0 to 27. Lower scores indicate better health scores and higher scores represent worse health status. Scores of 5, 10, 15, and 20 represent cutoffs for mild, moderate, moderately severe and severe depression, respectively.
Change in participant Generalized Anxiety Disorder (GAD-7) scores before and after interventions. | Each participant will be assessed at baseline (Day 1) and after the inpatient intervention (approximately Day 3 - 21) and at baseline (Day 1) and after the follow-up remote interventions (approximately 8 weeks after discharge).
  Change in anxiety level will be calculated using the GAD-7 questionnaire responses. The GAD-7 is a 7-items questionnaire with scores ranging from 0 to 21. Scores of 5, 10, and 15 represent cut-offs for mild, moderate, and severe anxiety, respectively.
Change in EEG spike frequency before, during, and after the intervention while participant is admitted to the DHMC epilepsy inpatient service. | Each participant will be assessed at baseline (Day 1) and after the inpatient intervention (approximately Day 3 - 21) and at baseline (Day 1) and after the follow-up remote interventions (approximately 8 weeks after discharge).
  EEG spike frequency will be determined by automated spike detection software
Change in seizure frequency from baseline to end of follow-up | Each participant will be assessed at baseline (Day 1) and after the inpatient intervention (approximately Day 3 - 21) and at baseline (Day 1) and after the follow-up remote interventions (approximately 8 weeks after discharge).
  Comparison of seizure data at baseline and post-interventions based on patient report of baseline and seizure calendar reporting
Qualitative analysis to identify themes in the creative writing and visual art subject matter. | After the inpatient intervention (approximately Day 3 - 21) and after each follow-up remote intervention (approximately 8 weeks after discharge).
  Participants assigned to either the creative writer or to the visual artist will supply their creations for analysis. The creative writing subject matter will be analyzed using N-Vivo software. Visual art subject matter will be coded for thematic content manually.
Change in quality of life measures for participants ultimately diagnosed with non-epileptic seizures compared to those diagnosed with epileptic seizures. | Each participant will be assessed at baseline (Day 1) and after the inpatient intervention (approximately Day 3 - 21) and at baseline (Day 1) and after the follow-up remote interventions (approximately 8 weeks after discharge).
  Change in quality of life for patients with non-epileptic seizures will be calculated using the QOLIE-10 questionnaire responses.The QOLIE-10 includes 10 questions. The score is calculated by the sum of scores for all questions divided by the number of items answered. Thus, if a patient skipped an item, it is not reflected in the total score. A lower score indicates a higher quality of life, and a higher score indicates a lower quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States